CLINICAL TRIAL: NCT00033007
Title: Motivational Incentives for Enhanced Drug Abuse Recovery: Drug Free Clinics
Brief Title: Motivational Incentives for Enhanced Drug Abuse Recovery: Drug Free Clinics - 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Maxine Stitzer, Ph.D., Johns Hopkins Bayview Medical Center
Organization: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: NIDA-CTN-0006-1; NCT00015405 (obsolete NCT alias)
Record Dates: First submitted 2002-04-05; First posted 2002-04-08 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2010-04

CONDITIONS: Substance-Related Disorders
Keywords: substance use disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Behavior Therapy

SUMMARY:
The purpose of this study is to test the utilization of incentive values (considerably lower than those typically used in research clinics) to motivate clients to attend treatment and initiate and sustain abstinence.

DETAILED DESCRIPTION:
The purpose of the proposed research is to implement and systematically evaluate, in community treatment settings, motivational incentive procedures that have been well researched and have proven efficacious in a variety of treatment research clinics.

ELIGIBILITY:
Inclusion Criterea:

* New intake to a drug-free CTP
* Evidence of cocaine or methamphetamine use, any reported use in past 2 weeks or positive urine screen at study intake. For those exiting a controlled environment, any stimulant use within two weeks of entering the controlled environment

Exclusion Criteria:

* Unable to give informed consent (fails simple consent quiz)
* Answers yes to question: Are you in recovery from gambling? That is, have you stopped gambling because of previous problems with gambling?

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 440
Dates: Start 2001-04; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
ASI
Cocaine use
AIDS risk behavior

CONTACTS AND LOCATIONS:
Overall Officials: Maxine Stitzer, Ph.D., Principal Investigator — Johns Hopkins University
Locations (11):
- United States (11):
  - MATRIX/LA Addictions Research, Los Angeles, California
  - Crossroads Managed Care Systems - Alamosa, Alamosa, Colorado
  - Arapahoe/Douglas Mental Health Network, Littleton, Colorado
  - Crossroads Managed Care Systems - Pueblo, Pueblo, Colorado
  - Crossroads Managed Care Systems - Trinidad, Trinidad, Colorado
  - LMG Programs, Inc., Stamford, Connecticut
  - Harbel Prevention and Recovery Center, Baltimore, Maryland
  - Thomas Jefferson Intensive Sub. Abuse TP, Philadelphia, Pennsylvania
  - Charleston Center, Charleston, South Carolina
  - Circle Park Behavioral Health Services - Florence, Florence, South Carolina
  - Circle Park Behavioral Health Services - Lake City, Florence, South Carolina

REFERENCES:
- See also: Data Elements — http://www.ctndatashare.org/protocol-ctndatashare/new-protocols/nida-ctn-0006